CLINICAL TRIAL: NCT02075060
Title: Evaluation of Immediate Preoperative Instillation (IPOI) of Mitomycin C Compared to Early Postoperative Instillation (IPOP) in Non-muscle Invasive Bladder Cancer
Acronym: IPOI vs IPOP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPOI vs IPOP
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Non Muscle-invasive Bladder Cancer
Keywords: low-grade; NMIBC
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPOI (Experimental): One arm with pre-operative instillation of mitomycine 1h before TURB (IPOI : Instillation pré-opératoire immédiate),
  Interventions: Procedure: IPOI (pre-operative)
- IPOP (Active Comparator): One arm with early post-operative instillation of mitomycine within 24 hours (IPOP : Instillation Post Opératoire Précoce).
  Interventions: Procedure: IPOP (post-operative)

INTERVENTIONS:
Procedure: IPOI (pre-operative)
  Arms: IPOI
Procedure: IPOP (post-operative)
  Arms: IPOP

SUMMARY:
The aim of this pilot study is to assess the efficacy and toxicity of immediate pre-operative instillation of mitomycin C compared to the standard early post-operative .

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Primary or recurrent bladder tumor with endoscopic papillary aspect,
* One or two bladder tumors,
* Cytology before TURB showing no high-grade cells,
* Patients without tutorship or subordination (ou curatorship),
* Patients under the general social security system or qualifying through a third party,
* Informed consent signed by the patient after clear and fair information.

Exclusion Criteria:

* Age < 18 years,
* Allergy to mitomycin C,
* Traumatic stenting,
* Upper tract urothelial cancer,
* Urethral invasion,
* History of muscle invasive bladder cancer,
* Extensive tumor (3 cm or more),
* Any contraindication to TURB,
* Simultaneous participation in another clinical research study,
* Patients not insured by the social security or not qualifying through a third party,
* Patients with enhanced protection, namely pregnant or lactating women, persons deprived of their liberty by a judicial or administrative decision, people staying in a health or social institution, adults under legal protection, and finally patients in emergency situations,
* Pregnant or lactating females or women of childbearing potential not willing to use an adequate method of birth control for the duration of the study (i.e. hormonal / mechanical contraceptive : oral, injectable, transdermal, implantable, intrauterine or surgical device: tubal ligation, hysterectomy, total oophorectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-01-18 (Estimated); Study Completion 2018-01-18 (Estimated)

PRIMARY OUTCOMES:
PFS | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques IRANI, MD, PhD, Principal Investigator — Poitiers University Hospital
Locations (3):
- France (3):
  - Bicêtre Hospital, Le Kremlin-Bicêtre
  - Poitiers University Hospital, Poitiers
  - Rouen University Hospital, Rouen